CLINICAL TRIAL: NCT05887063
Title: Investigating the Feasibility, Acceptability, and Impact of an Online UK Dementia Awareness Course for Informal Caregivers: A Mixed Methods Study
Brief Title: Trialling an Online UK Dementia Awareness for Caregivers Course
Acronym: DAC-UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22375.001
Record Dates: First submitted 2023-05-05; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Dementia; Caregiver Burden
Keywords: Dementia; Caregiver; Intervention; Biopsychosocial
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dementia Awareness Course (Experimental): Participants attended one half-day Dementia Awareness course as a part of a group, delivered online
  Interventions: Other: Dementia Awareness Course UK
- Treatment as Usual (No Intervention): Participants did not receive any active treatment but were able to access their usual supports

INTERVENTIONS:
Other: Dementia Awareness Course UK — An online course delivered to a small group of informal caregivers in between 3 and 4 hours. The course is made up of three modules: what is dementia, positive engagement and caring for someone with dementia. The course is delivered by one facilitator and includes teaching, discussions and activities.
  Arms: Dementia Awareness Course

SUMMARY:
The purpose of this study is to investigate whether an online Dementia Awareness Course is feasible for delivery and acceptable to informal caregivers of people living with dementia in the UK. It will also explore the impact of the course on different caregiver outcomes.

DETAILED DESCRIPTION:
All participants were given information on the study before providing informed consent. The participants were screened against eligibility criteria before being randomly allocated to either the treatment condition of attending the course, or the control condition of treatment as usual. Participants completed 5 outcome measures and a demographics questionnaire at baseline. The treatment group then attended a one-off half-day Dementia Awareness Course online, delivered by one trainee clinical psychologist. A month later, all participants completed the same 5 outcome measures and those who attended the course also attended a one-to-one half an hour online semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified informal caregiver of a person living with dementia in the community.
* Residing in the U.K.
* Ability to engage in a course delivered in English
* Have access to an internet-connected device capable of videoconferencing (camera and microphone functioning)
* Available to attend pre-specified dates for DAC-UK delivery.

Exclusion Criteria:

* Person living with dementia residing in residential care
* Professional caregiver of people living with dementia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Percentage of target sample recruited within 6 months. | 6 months
  Feasibility of recruitment, considered feasible if full sample successfully recruited within 6 month time frame
Percentage of participants retained at follow-up to measure feasibility of the study design. | 1 month
  75% considered indicative of a feasible study design
Percentage of completion of outcome measures to measure feasibility and acceptability. | Baseline and 1 month
  75% considered indicative of feasible and acceptable outcome measures
Retention and attendance percentages to measure feasibility and acceptability of the intervention. | 1 month
  60% considered indicative of feasible and acceptable intervention
Qualitative acceptability of the intervention, as measured by qualitative thematic analysis of participant interviews to capture themes regarding participant experience of the course. | 1 month
  Exploratory thematic analysis

SECONDARY OUTCOMES:
Change from baseline in the mean Zarit burden inventory scores at one-month follow up | Baseline and 1 month
  Exploratory outcome measure - questionnaire. The short-form Zarit burden inventory (ZBI) is a 12-item questionnaire that measures caregiver's perceived burden as a result of their role. Each item is scored from 0 (never) to 4 (nearly always) where a low score is indicative of a low sense of burden. The ZBI is one of the most commonly used measures for burden in the field and has been shown to have high levels of validity and reliability.
Change from baseline in the mean Quality caregiver-patient relationship (QCPR) scores at one-month follow up | Baseline and 1 month
  Exploratory outcome measure - questionnaire. The carer version of the quality of the caregiver patient relationships (QCPR) is a 14-question survey that captures the positive and negative aspects of the caregiving relationship. The questions are scored on a 5-point Likert scale where 1 is totally disagree and 5 is totally agree. Six items are reversed scored (2, 3, 8, 10, 11, 13). A score of less than 42 is considered indicative of a poor caregiver-patient relationship, a score of 42-56 is labelled as a standard relationship, with scores of higher than 56 indicating a good relationship. Reliability and validity of the QCPR have been found to be high.
Change from baseline in the mean GAIN measure scores at one-month follow up | Baseline and 1 month
  Exploratory outcome measure - questionnaire. The gain in Alzheimer's care instrument (GAIN) comprises of 10 questions that cover the possible positive aspects of a caregiving role in terms of relationship with the person living with dementia, self-reflection and personal development. Each question is scored from 0 to 5 (disagree a lot to agree a lot) where a high score suggests a high level of positive gain from caregiving. This tool has been found to be valid and reliable for use.
Change from baseline in the mean approaches to dementia (ADQ-19) scores at one-month follow up | Baseline and 1 month
  Exploratory outcome measure - questionnaire. The approaches to dementia questionnaire (ADQ-19) is a 19-question survey that measures an individual's attitudes towards dementia and people living with dementia. Each question is scored on a five-point Likert scale from 0 (strongly agree) to 4 (strongly disagree). Reverse scoring is used on items 5, 7, 9, 11, 12, 15, 16, 17, 18, 19, and an overall high score indicates positive attitudes towards dementia and person living with dementia. The ADQ-19 has been shown to have good reliability (α=0.76 for hope, α=0.85 for person-centredness) and validity when compared with similar measures and qualitative observations.
Change from baseline in the mean short sense of competence (SSCQ) scores at one-month follow up | Baseline and 1 month
  Exploratory outcome measure - questionnaire. The short sense of competence questionnaire (SSCQ) is a 7-item questionnaire that measures an individual's sense of competence in their role as a caregiver. Each item is scored on a five-point Likert scale from 1 to 5, where 1 is agree strongly and 5 is disagree strongly. Scores can range from 7 to 35 with higher scores indicating a greater sense of competence/satisfaction. The SSCQ has been found to have high construct validity (r=0.88) when compared to the original sense of competence questionnaire and alongside this, high reliability (α=0.76).

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Spector, Principal Investigator — UCL
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stoner CR, Lakshminarayanan M, Mograbi DC, Vaitheswaran S, Bertrand E, Schimidt Brum P, Durgante H, Ferri CP, Mkenda S, Walker R, Dotchin C, Paddick SM, Chandra M, Krishna M, Du B, Shaji KS, Fisher E, Spector A. Development and acceptability of a brief, evidence-based Dementia Awareness for Caregivers course in low- and middle-income countries. Dementia (London). 2022 Feb;21(2):598-617. doi: 10.1177/14713012211055316. Epub 2021 Dec 9. PMID 34886707

DOCUMENTS (1):
  • Informed Consent Form (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05887063/ICF_000.pdf